CLINICAL TRIAL: NCT06655831
Title: Study on the Key Mechanisms of Abnormal T Cell Activation and Differentiation in IgG4-Related Ophthalmic Disease
Brief Title: Key Mechanisms of Abnormal T Cell Activation and Differentiation in IgG4-Related Ophthalmic Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SZZ1
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: IgG4-Related Diseases
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Lacrimal gland tissue samples from IgG4-ROD patients and patients with lacrimal gland ptosis undergoing surgical repositioning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IgG4-ROD: IgG4-ROD patients from the Department of Ophthalmology at Peking University Third Hospital.
- Lacrimal gland ptosis: Patients with lacrimal gland ptosis undergoing surgical repositioning fromthe Department of Ophthalmology at Peking University Third Hospital.

SUMMARY:
IgG4-related disease (IgG4-RD) is a newly recognized chronic inflammatory condition caused by immune system dysfunction. It is characterized by the infiltration of IgG4+ plasma cells, dense fibrosis, and inflammation involving veins and eosinophils. Common symptoms include elevated serum IgG4 levels and the formation of tumor-like growths that can affect almost any organ, leading to pressure on tissues, irreversible damage, and even organ failure. While estimates suggest a prevalence of 0.28 to 1.08 per 100,000 people, this might be an underestimation due to limited awareness, the new definition of the disease, and its subtle onset.

IgG4-related ophthalmic disease (IgG4-ROD) is a subtype of IgG4-RD that affects the eye area, particularly the lacrimal glands, extraocular muscles, and surrounding nerves. It often presents as painless swelling of the lacrimal glands in one or both eyes, sometimes with discomfort or a sensation of a foreign body. It can also cause thickening of eye muscles, leading to symptoms like bulging eyes, blurred vision, or double vision. In some cases, mass lesions in the orbit may press on the optic nerve, potentially leading to permanent vision loss. While there is currently no cure for IgG4-ROD, steroids are used as the main treatment to control inflammation and fibrosis. However, the disease often recurs, with recurrence rates for IgG4-RD reported between 24% and 63% in various studies. Understanding the causes of IgG4-ROD could help develop better treatments and reduce the chances of relapse.

Studies suggest that T cells play a key role in the development of IgG4-RD, including IgG4-ROD. CD4+ T cells are the main immune cells found in affected tissues. They can help B cells multiply and produce IgG4 antibodies and contribute to tissue fibrosis by releasing certain signaling molecules. Despite treatment with rituximab, a drug that targets B cells, many IgG4-RD patients experience relapses, indicating that T cells remain important in driving the disease. Among the T cell subtypes, T follicular helper cells (Tfh) and CD4+ cytotoxic T cells (CD4+ CTLs) are particularly relevant. Tfh cells support B cells in producing IgG4 antibodies, while CD4+ CTLs can contribute to tissue fibrosis by releasing factors like TGF-β, IL-1β, and IFN-γ. However, the detailed mechanisms of how T cells become abnormally activated and differentiated in IgG4-ROD remain unclear.

This study will use samples from the lacrimal glands, blood, and tears of IgG4-ROD patients to investigate how T cells become abnormally active and differentiate in this condition. The findings could identify new targets for therapy, helping to reduce the recurrence of IgG4-ROD and provide insights into treating other forms of IgG4-RD.

DETAILED DESCRIPTION:
Immunoglobulin-G4 related disease (IgG4-RD) is a newly defined immune-mediated chronic inflammatory disease with fibrosis, characterized by lymphoplasmacytic infiltration predominantly consisting of IgG4+ plasma cells, along with storiform fibrosis, obliterative phlebitis, and eosinophil infiltration. The most common clinical manifestations of IgG4-RD include significantly elevated serum IgG4 levels and mass-like lesions, which can affect nearly any part of the body, leading to compression and irreversible damage to affected organs and surrounding tissues, potentially resulting in organ failure. Despite reports estimating the prevalence of IgG4-RD to be between (0.28~1.08)/100,000, the actual prevalence might be higher due to its recent definition, limited awareness among clinicians and patients, and its insidious onset.

Immunoglobulin-G4 related ophthalmic disease (IgG4-ROD) refers to IgG4-RD mass-like lesions involving the lacrimal gland, extraocular muscles, supraorbital nerve, infraorbital nerve, and other orbital structures, leading to orbital lesions. Among these, lacrimal gland involvement is the most common, manifesting as painless, unilateral or bilateral swelling, sometimes accompanied by foreign body sensation or eye discomfort. Extraocular muscle involvement can present as muscle enlargement, potentially causing proptosis, blurred vision, and diplopia in severe cases. Orbital mass lesions may also compress the optic nerve, leading to irreversible vision loss. While there is currently no cure for IgG4-ROD, glucocorticoids are used as the first-line treatment to control inflammation and fibrosis associated with the mass-like lesions. IgG4-ROD is prone to relapse, and though there are no studies specifically on its recurrence rate, different studies have reported relapse rates of IgG4-RD patients during follow-up ranging from 24% to 63%. The exact etiology and pathogenesis of IgG4-ROD remain unclear, and further elucidation of these aspects would facilitate the identification of new therapeutic targets, reduce relapse rates, and potentially achieve a cure.

Multiple studies on various forms of IgG4-RD suggest a critical role of T cells in the pathogenesis of IgG4-RD, including IgG4-ROD. First, CD4+ T cells constitute the majority of infiltrating lymphocytes in the lesions of IgG4-RD. These CD4+ T cells induce B cell proliferation and class-switching through cytokine secretion and contribute to tissue fibrosis. Additionally, IgG4-RD patients treated with rituximab exhibit high relapse rates, with post-relapse B cell clones expanding differently compared to pre-treatment . This evidence strongly supports the central role of T cells in IgG4-RD. Among the T cell subpopulations implicated in IgG4-RD pathogenesis, T follicular helper cells (Tfh) and CD4+ cytotoxic T lymphocytes (CD4+ CTLs) are particularly notable. Tfh cells promote ectopic germinal center formation and B cell class-switching to IgG4+ plasma cells through IL-21 secretion, while CD4+ CTLs contribute to tissue fibrosis by secreting TGF-β, IL-1β, and IFN-γ . However, the mechanisms underlying abnormal T cell activation and differentiation in both IgG4-ROD and other IgG4-RD remain poorly understood.

This study aims to investigate key pathways involved in abnormal T cell activation and differentiation in IgG4-ROD by conducting a series of in vitro experiments using surgical tissue samples, peripheral blood, and tear fluid from patients with IgG4-ROD. These experiments include RNA sequencing (RNA-Seq), enzyme-linked immunosorbent assays (ELISA), and in vitro cell co-culture. The goal is to identify critical pathways in the pathogenesis of IgG4-ROD and to clarify their roles in the disease process, providing new therapeutic targets to reduce the recurrence rate of IgG4-ROD. This research may also offer insights into the mechanisms and treatment of other IgG4-related diseases.

Study Population

This study involves patients from the Department of Ophthalmology at Peking University Third Hospital, including lacrimal gland tissue samples from IgG4-ROD patients (experimental group) and patients with lacrimal gland ptosis undergoing surgical repositioning (control group). The inclusion and exclusion criteria are as follows:

Inclusion Criteria

Experimental Group: IgG4-ROD patients with lacrimal gland involvement, diagnosed based on 2014 and 2020 Japanese criteria for IgG4-ROD and IgG4-RD:

Clinical and imaging features: characteristic diffuse or localized swelling or nodular formations of the lacrimal glands.

Serological diagnosis: Elevated serum IgG4 concentration (>135 mg/dL).

Histopathological diagnosis (meeting 2 of the 3 criteria below):

Dense lymphoplasmacytic infiltration with fibrosis. IgG4+ plasma cell/IgG+ plasma cell ratio >40%, and >10 IgG4+ plasma cells per high-power field.

Characteristic fibrosis, especially storiform fibrosis, or obliterative phlebitis.

Control Group: Patients with lacrimal gland ptosis confirmed by pathology and clinical/imaging features, requiring surgical repositioning.

Exclusion Criteria

Presence of other autoimmune diseases like Sjögren's syndrome, systemic lupus erythematosus, or rheumatoid arthritis.

Lacrimal gland pathology indicating other orbital diseases such as MALT lymphoma or inflammatory pseudotumor.

Other exclusion criteria include mental disorders, malignancies, or any condition deemed unsuitable for study participation.

Study Methods

Collection of Clinical Information Patient demographics, medical history, and necessary diagnostic test results (e.g., imaging, serum IgG levels) are recorded. Ocular examinations include visual acuity, intraocular pressure, Ocular Surface Disease Index (OSDI), corneal fluorescein staining (CFS), tear film break-up time (FBUT), and Schirmer's test, among others.

Collection of Samples Tear fluid (about 15 µL per eye) is collected using a capillary tube and stored at -80°C. A portion (50-100 mg) of the resected lacrimal gland tissue is reserved for this study, while the rest is used for pathological analysis. Blood samples (approximately 10 mL) are drawn for preparing peripheral blood mononuclear cells (PBMCs).

Bulk RNA-Seq Analysis of Lacrimal Gland Tissue Total RNA is extracted from lacrimal gland tissue using the Trizol method, followed by RNA quality assessment with an Agilent bioanalyzer. A cDNA library is constructed and sequenced using Illumina technology. Data processing includes quality control with fastp, alignment using HISAT2, and gene expression quantification with featureCounts. Differential expression analysis is performed using DESeq2, and Gene Set Enrichment Analysis (GSEA) is conducted. Immune cell composition in the tissue is analyzed using xCell and CIBERSORTx.

Enzyme-linked Immunosorbent Assay (ELISA) ELISA is used to analyze key pathways identified in the RNA-Seq results, using specific kits according to the manufacturer's instructions.

In Vitro Co-culture Experiments An in vitro co-culture system of IgG4-ROD patient lacrimal gland cells and PBMCs is established to simulate the immune microenvironment of the lacrimal gland. Based on RNA-Seq and ELISA results, targeted interventions are applied to this system. IgG4/IgG1 ratios in the supernatant serve as an indicator, with higher values suggesting stronger pathogenic effects.

ELIGIBILITY:
Inclusion Criteria:

* Experimental Group: IgG4-ROD patients with lacrimal gland involvement, diagnosed based on 2014 and 2020 Japanese criteria for IgG4-ROD and IgG4-RD:

Clinical and imaging features: characteristic diffuse or localized swelling or nodular formations of the lacrimal glands.

Serological diagnosis: Elevated serum IgG4 concentration (>135 mg/dL).

Histopathological diagnosis (meeting 2 of the 3 criteria below):

Dense lymphoplasmacytic infiltration with fibrosis. IgG4+ plasma cell/IgG+ plasma cell ratio >40%, and >10 IgG4+ plasma cells per high-power field.

Characteristic fibrosis, especially storiform fibrosis, or obliterative phlebitis.

Control Group: Patients with lacrimal gland ptosis confirmed by pathology and clinical/imaging features, requiring surgical repositioning.

Exclusion Criteria:

* Presence of other autoimmune diseases like Sjögren's syndrome, systemic lupus erythematosus, or rheumatoid arthritis.

Lacrimal gland pathology indicating other orbital diseases such as MALT lymphoma or inflammatory pseudotumor.

Other exclusion criteria include mental disorders, malignancies, or any condition deemed unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patients from the Department of Ophthalmology at Peking University Third Hospital, including lacrimal gland tissue samples from IgG4-ROD patients (experimental group) and patients with lacrimal gland ptosis undergoing surgical repositioning (control group).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Bulk RNA-Seq Analysis of Lacrimal Gland Tissue | At the time of enrollment.
  Total RNA is extracted from lacrimal gland tissue using the Trizol method, followed by RNA quality assessment with an Agilent bioanalyzer. A cDNA library is constructed and sequenced using Illumina technology. Data processing includes quality control with fastp, alignment using HISAT2, and gene expression quantification with featureCounts. Differential expression analysis is performed using DESeq2, and Gene Set Enrichment Analysis (GSEA) is conducted. Immune cell composition in the tissue is analyzed using xCell and CIBERSORTx.

SECONDARY OUTCOMES:
Enzyme-linked Immunosorbent Assay (ELISA) | At the time of enrollment.
  ELISA is used to analyze key pathways identified in the RNA-Seq results, using specific kits according to the manufacturer's instructions.
In Vitro Co-culture Experiments | At the time of enrollment.
  An in vitro co-culture system of IgG4-ROD patient lacrimal gland cells and PBMCs is established to simulate the immune microenvironment of the lacrimal gland. Based on RNA-Seq and ELISA results, targeted interventions are applied to this system. IgG4/IgG1 ratios in the supernatant serve as an indicator, with higher values suggesting stronger pathogenic effects.